CLINICAL TRIAL: NCT03567369
Title: Comparative Study of the Preoperative Efficacy of Traumeel Versus Dexamethasone in Control of Pain, Swelling and Trismus After Mandibular Third Molar Extractions
Brief Title: 92/5000 Preoperative Efficacy of Traumeel Versus Dexamethasone in the Control of Pain, Swelling and Trismus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Federal University of the Valleys of Jequitinhonha and Mucuri (Other)
Responsible Party: Principal Investigator, Marcos Luciano Pimenta Pinheiro, Principal Investigator, Federal University of the Valleys of Jequitinhonha and Mucuri
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 24042018
Record Dates: First submitted 2018-05-14; First posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-05

CONDITIONS: Molar, Third; Surgery
Keywords: Third molar; Surgery; Swelling
MeSH Terms: interventions — Dexamethasone; dexamethasone acetate; Calcium Dobesilate; Traumeel S

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Experimental): Dexamethasone 4,0 mg / mL
  Interventions: Drug: Dexamethasone
- Traumeel S (Experimental): Traumeel 2,2 mg / mL
  Interventions: Drug: Traumeel S

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 4,0 mg/mL
  Other Names: Dexamethasone Acetate; Decadron®
  Arms: Dexamethasone
Drug: Traumeel S — Traummel S 2,2 mg/mL
  Arms: Traumeel S

SUMMARY:
To compare the efficacy of intramuscular injection of two anti-inflammatory drugs, Traumeel and Dexamethasone, used in the control of postoperative complications pain, edema and trismus after third molar extraction mandibular

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication of asymptomatic bilateral extractions of lower third molars;
* Aged 18 years or older;
* Have a good health and no disease.

Exclusion Criteria:

• Patients with history of any medication treatment within 15 days before the beginning of the research, history of allergy to the drugs, substances or materials used in this study, pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative sequelae following thir molar extraction | up to seven days postoperative
  During the postoperative intervals of 24, 48 and 72 hours and seven days, the swelling was determined using linear measures in the face and trismus by maximum mouth opening. The postoperative pain was self-recorded by the patient using visual analogue scale in 72 hours with an interval of eight hours

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal dos Vales do Jequitinhonha e Mucuri, Diamantina, Minas Gerais, Brazil